CLINICAL TRIAL: NCT05431569
Title: A Phase IIa Study to Evaluate the Efficacy and Safety of 6MW3211 in Patients With Advanced Lung Cancer Who Had Failed Therapy With PD-1/L1 Inhibitor
Brief Title: A Phase IIa Study to Evaluate the Efficacy and Safety of 6MW3211 in Patients With Advanced Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6MW3211-2022-CP203
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Advanced Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6MW3211 (Experimental): 6MW3211injection,30mg/kg,Q2W
  Interventions: Drug: 6MW3211

INTERVENTIONS:
Drug: 6MW3211 — 6MW3211 injection ,30mg/kg,iv drip，Q2W
  Other Names: 6MW3211injection

SUMMARY:
A non-randomized, open, Simon'soptimal2-stage study to evaluate the efficacy and safety of 6MW3211 in patients with advanced Lung Cancer who had failed therapy with PD-1/L1 Inhibitor.

DETAILED DESCRIPTION:
36 to 64 patients with advanced lung cancer who failed pD-1 /L1 inhibitor treatment will be inrolled.

Cohort 1:20 to 33 patients with non-small cell lung cancer (NSCLC) Cohort 2:16 to 31 patients with small cell lung cancer (SCLC)

ELIGIBILITY:
Inclusion Criteria:

1. years≥18
2. cohort1：Locally advanced or metastatic NSCLC (stage IIIB-IV) confirmed by histological or cytological evidence that cannot be treated with radical surgical resection and cannot be treated with radical synchronous/sequential chemoradiotherapy.

cohort2:Extensive stage small cell lung cancer (ES-SCLC) confirmed byhistologically or cytologically 3.Patients who had failed therapy with PD-1/L1 Inhibitor. 4.≥5 slides of unstained tumor tissue should be provided 5.EGFR, ALK, ROS1 were negative 6.ECOG 0 or 1 7.At least one extracranial measurable target evaluated by RECIST1.1 8.Expected survival≥3 months 9.Suitable organs and hematopoietic functions 10.Women and men of reproductive age must agree to use effective contraception from the date of signing the informed consent until 6 months after the last administration of 6MW3211 injection, and women of reproductive age must have negative serum pregnancy test results within 7 days prior to administration.

11.Sign informed consent voluntarily

-

Exclusion Criteria:

1. Patients who had received immunotherapy other than pD-1 /L1 inhibitors
2. Patients who were discontinued due to grade ≥3 serious immune-related adverse events (irAE) when treated with a PD-1/L1 inhibitor
3. Patients who had received anti-PD-1 /L1 inhibitor,have had immune pneumonia or immune myocarditis
4. Patients who had malignant tumors other than NSCLC or SCLC within 5 years
5. Patients with active central nervous system (CNS) metastasis or meningeal metastasis.
6. Adverse reactions related to previous treatments failed to recover to CTCAE 5.0 ≤1
7. patients with autoimmune diseases that are likely to recur
8. Patients with history of interstitial lung disease or have non-infectious pneumonia
9. Uncontrolled systemic diseases after treatment.
10. Patients with active tuberculosis
11. Patients with severe infection or requiring antibiotic treatment within the first 4 weeks prior to initial administration
12. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage
13. Prior blood transfusion or hematopoietic stimulator therapy within 4 weeks prior to initial dosing
14. Patients who have previously received antitumor therapy
15. Patients requiring systemic glucocorticoids or other immunosuppressive agents within 14 days prior to initial dosing or during the study period
16. Patients who were allergic to any composition of investigational drug
17. Patients with chronic active hepatitis B or active hepatitis C
18. Patients who received other investigational drugs within 4 weeks prior to initial dosing
19. Patients who underwent major surgery within 30 days prior to first administration
20. History of drug or substance abuse in the past 1 year
21. Live vaccine was administered within 30 days prior to first administration
22. Have the history of neuropsychiatric disorders
23. Women who are pregnant or breastfeeding
24. Patients had other factors that might have forced them to terminate the study by investigator's judgment -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24mouths or intolerable toxicity, disease progression or death, patient withdrawal of informed consent, withdrawal from the study and so on
  The percentage of (PR+CR) after treatment to the total number of cases was calculated

IPD SHARING:
Plan to Share IPD: No